CLINICAL TRIAL: NCT06843512
Title: Exploring the Influence of GLP-1 Medication on Food Attitudes and Selection in a Virtual Reality Buffet
Brief Title: Identifying Changes in Food Behaviors Associated With Beginning GLP-1 Medication
Status: Recruiting | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Travis Masterson, Assistant Professor and Director of the Health, Ingestive Behavior, and Technology Lab, Penn State University
Other Study IDs: STUDY00026642
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Weight Loss; Food Selection
Keywords: GLP-1; Weight Loss; Virtual Reality; Food behavior
MeSH Terms: conditions — Weight Loss; Food Preferences

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Other: GLP-1 Medication Initiation — One visit before starting GLP-1 medication and one visit 3 months after. No other changes administered between visits.

SUMMARY:
In recent years, GLP-1 medications have become a widely employed approach by physicians to address weight concerns in patients and lead to weight loss. Little is known, however, about how these medications may alter an individual's attitude towards food, food reactivity, or the specific types and amounts of foods an individual will choose. The purpose of this study is to observe the changes an individual experiences in their relationship and reaction to food and in their food selection prior to or within the first two weeks of taking GLP-1 medication to after three months on the medication. The researchers of this study believe that an understanding of such changes can inform questions seeking to ensure maintenance of appropriate nutrient balance within individuals on weight loss medications.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+) with overweight or obesity (BMI >25 kg/m2)
* Not currently taking an incretin-based medication at baseline
* Recently (within two weeks) prescribed a GLP-1, can be included if they have a obesity-related co-occurring condition (diabetes, hypertension, cardiovascular disease, dyslipidemia)
* Have had no prior diagnosis of cognitive or physical disability, dyslexia, or epilepsy.
* Fluent in English

Exclusion Criteria:

* Adults (18+) without overweight or obesity
* <18 years of age at time of testing
* Adults not taking a GLP-1 Medication
* Adults taking a compound GLP-1
* Adults on GLP-1 medication for longer than 2 weeks at baseline
* Have had a prior diagnosis of cognitive or physical disability, dyslexia, or epilepsy.
* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from a list of medical patients prescribed GLP-1 medication by their physicians (located in offices near State College or Hershey, PA) and who volunteered to be contacted regarding studies they are eligible for.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Total Weight of Food Selected in the VR Buffet at 3 Months | Baseline and 3 months
Change from Baseline in Total Calories of Food Selected in the VR Buffet at 3 Months | Baseline and 3 months
Change from Baseline in Energy Density of Food Selected in the VR Buffet at 3 Months | Baseline and 3 months
Change from Baseline in Variety of Food Selected in the VR Buffet at 3 Months | Baseline and 3 months

SECONDARY OUTCOMES:
Change in Baseline Weight Watchers Food Noise Score at 3 Months | Baseline and 3 months
  Based on participant's answers to the WW Food Noise questionnaire; Scale of 1-5, 1 being strongly disagree and 5 being strongly agree; Higher scores mean more food noise
Change in Baseline 9-question External Food Cue Responsiveness Questionnaire Score at 3 Months | Baseline and 3 months
  Answers are on a 1-4 scale with 1 being "Rarely" and 4 being "A lot"; higher scores suggest more external food cue reactivity
Change in Baseline Adult Eating Behavior Score at 3 Months | Baseline and 3 months
  Answers on a 1-5 scale with 1 being "Strongly disagree" and 5 being "Strongly agree"; 8 subscales, high scores indicate greater expression of subscale measure
Change in Baseline Three-Factor Eating Questionnaire Score at 3 Months | Baseline and 3 months
  Rated on a scale of 1-4 with 1 being "Definitely false" and 4 being "Definitely true"; 3 subscales, higher scales on each means greater expression of that behavior
Change in Baseline General Food Craving-Trait Scale Score at 3 Months | Baseline and 3 months
  Rated on a 0-5 scale with 0 being "Never/not applicable" and 5 being "Always"; higher scores mean more food dependent
Change in Baseline Buffet Food Liking Scores at 3 Months | Baseline and 3 months
  Rated on a 0-100 scale with 0 being "Dislike extremely" and 100 being "Like extremely"; high scores mean greater liking of the food

OTHER OUTCOMES:
Change in Baseline BMI at 3 Months | Baseline and 3 months
  Calculated from height and weight collected at the end of both sessions

CONTACTS AND LOCATIONS:
Overall Officials: Travis Masterson, Principal Investigator — The Pennsylvania State University
Locations (1):
- Health, Ingestive Behavior, and Technology Laboratory of Pennsylvania State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No